CLINICAL TRIAL: NCT02464358
Title: The Impact of an Information-Motivation-Behavioral Skills (IMB) Based Educational Intervention to Improve Gardasil Use in a Population of Undergraduate Women
Brief Title: An Information-Motivation-Behavioral Skills (IMB) Intervention to Promote Human Papillomavirus Vaccination Among Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Dean Cruess, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H11-272
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMB Intervention Group (Experimental): The IMB group received an HPV Vaccination Information Statement (VIS) often given to individuals prior to vaccination. In addition, they received the following:
  1. Additional educational content related to HPV, Cervical Cancer, and HPV vaccination,
  2. Motivational content to help identify and problem-solve benefits and barriers to vaccination,
  3. Skills-building content, including brief communication skills training and ways to access the vaccine.
  Interventions: Behavioral: IMB Intervention Group
- Attention Control Group (Active Comparator): The attention control group also received an HPV Vaccination Information Statement (VIS) often given to individuals prior to vaccination. In addition, to maintain consistency with the treatment's presentation format, participants watched a set of short video clips encompassing aspects of women's general and sexual health.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: IMB Intervention Group — Participants in the IMB group received information specific to HPV, cervical cancer, and the HPV vaccine. This information was delivered in a group setting, and it was delivered via a PowerPoint presentation that included short video clips.
  Other Names: IMB Based Educational Program
  Arms: IMB Intervention Group
Behavioral: Attention Control — Participants in the attention control arm watched a PowerPoint that contained a series of short video clips encompassing aspects of women's general and sexual health. This was also conducted in a group setting.
  Arms: Attention Control Group

SUMMARY:
HPV infections are prominent among college-aged women. Although HPV vaccines decrease women's risk for cervical cancer, vaccination rates remain inadequate. This study explored the utility of an Information-Motivation-Behavioral Skills intervention in promoting HPV vaccination knowledge, motivation, and behavioral skills among college aged women.

DETAILED DESCRIPTION:
HPV infections are prominent among college-aged women. Although HPV vaccines decrease women's risk for cervical cancer, vaccination rates remain inadequate. This study explored the utility of an Information-Motivation-Behavioral Skills intervention in promoting HPV vaccination knowledge, motivation, and behavioral skills among college aged women.

Methods: Participants were randomly assigned to a single-session intervention or attention-control arm and were assessed at pre-intervention, post-intervention, and at 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a psychology course at the University of Connecticut

Exclusion Criteria:

* Completion of the HPV vaccination series

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
HPV, Cervical Cancer, and HPV Vaccine Knowledge Questionnaire | One month
  Consistent with studies based on the IMB model,, participants were assessed on their level of knowledge regarding information about HPV, the HPV vaccine, and cervical cancer.
Vaccination Motivation Questionnaire | One month
  Consistent with studies based on the IMB model, motivation to get vaccinated was assessed through five questionnaires to measure different aspects of motivation: perceived motivation, attitudes related to getting vaccinated, perceived social norms to getting vaccinated, behavioral intentions, and perceived risk for HPV/cervical cancer.
Behavioral Skills Questionnaire | One Month
  Consistent with studies based on the IMB model, participants' belief and confidence in their ability to get vaccinated were assessed with questions adapted from these studies.

SECONDARY OUTCOMES:
Behavioral uptake of the HPV vaccine Questionnaire | One month

CONTACTS AND LOCATIONS:
Overall Officials: Dean G Cruess, Ph.D., Principal Investigator — University of Connecticut; Giselle K Perez, Ph.D., Study Director — Massachusetts General Hospital